CLINICAL TRIAL: NCT04196101
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study of EDP-938 Administered Orally for the Treatment of Acute Upper Respiratory Tract Infection With Respiratory Syncytial Virus in Ambulatory Adult Subjects (RSVP)
Brief Title: A Study to Assess EDP-938 for the Treatment of Acute Upper Respiratory Tract Infection With Respiratory Syncytial Virus in Adult Subjects
Acronym: RSVP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDP 938-102
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Syncytial Virus
Keywords: RSV
MeSH Terms: interventions — EDP-938

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP-938 (Experimental): Subjects will take EDP-938 tablets (800 mg) once a day orally for 5 days
  Interventions: Drug: EDP-938
- Placebo (Placebo Comparator): Subjects will take EDP-938 matching placebo tablets once a day orally for 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-938 — Four tablets daily for 5 days
  Arms: EDP-938
Drug: Placebo — Four tablets daily for 5 days
  Arms: Placebo

SUMMARY:
This was a randomized, double-blind, placebo-controlled, multicentre, phase 2 study to evaluate the efficacy, safety and tolerability of orally administered EDP-938 in adults with RSV infection.

DETAILED DESCRIPTION:
Subjects (aged 18 to 75 years, inclusive) with up to 48 hours of upper respiratory tract infection (URTI) symptoms who tested positive for respiratory syncytial virus (RSV) and negative for influenza virus by rapid testing (ie, Rapid Viral Screen). Subjects with stable asthma or chronic obstructive pulmonary disease (COPD) were allowed in the study.

Eighty-two (82) subjects were enrolled in this Phase 2b, randomized, double-blind, placebo-controlled, multicentre study of EDP-938 administered orally for the treatment of acute URTI with confirmed RSV infection in ambulatory adult subjects.

For each subject, the duration of study participation was approximately 2 weeks and consisted of 3 periods: Screening (occurs on Day1), Treatment (5 days), and Follow-up (9 days after last dose).

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document must be signed and dated by the subject
* Male or female individuals aged 18 to 75 years, inclusive.
* Up to 48 hours of URTI symptoms with at least one of the following symptoms:

Nasal discharge, nasal congestion, malaise/tiredness, headache, sinus congestion, sneezing, sore throat, hoarseness, cough, shortness of breath, respiratory wheeze, earache, and/or symptoms of fever.

* Positive for RSV infection and negative for influenza virus based on rapid diagnostic.
* Must be willing and able to adhere to the study assessments, visit schedules, prohibitions, and restrictions, as described in this protocol.

Exclusion Criteria:

* SARS-CoV-2 positive within 28 days of Screening or at Screening following signature of full ICF.
* Clinical evidence of a lower respiratory tract infection, as determined by the Investigator.
* Anticipated need for hospitalization or emergency room care within 24 hours of Screening.
* Receipt of systemic antiviral, antibacterial, antifungal, or antimycobacterial therapy within 7 days of Screening and for the duration of the study
* Awareness of concomitant respiratory infections that are viral (other than RSV), bacterial, or fungal, including systemic bacterial or fungal infections, within 7 days of Screening.
* Frailty scale score ≥4 at Screening.
* History of chronic liver disease (eg, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, autoimmune hepatitis, nonalcoholic steatohepatitis, and/or alcoholic liver disease); a history of biliary disease (eg, primary sclerosing cholangitis, cholecystitis, choledocholithiasis); or a history of portal hypertension. A diagnosis of hepatic steatosis (fatty liver) is not exclusionary.
* Heart disease: any congenital heart disease, acute or chronic heart failure, ischemic heart disease, congenital long QT syndrome, or any clinical manifestation resulting in QT interval prolongation.
* Neurological and neurodevelopmental disorders (including disorders of the brain, spinal cord, peripheral nerve, and muscle, eg, cerebral palsy, epilepsy [seizure disorders], stroke, muscular dystrophy, or spinal cord injury).
* Malignant tumor or history of malignancy that may interfere with the aims of the study or a subject completing the study.
* Prior receipt or the subject is waiting to receive a bone marrow, stem cell, or solid organ transplantation.
* Diagnosis of cystic fibrosis.
* Known positive human immunodeficiency virus, active hepatitis A virus infection, chronic hepatitis B virus infection, and/or current or treated hepatitis C virus infection.
* Prior or planned ileal resection or bariatric surgery.
* Pregnant or nursing female subjects.
* History of alcohol addiction or current heavy alcohol use defined as: >14 standard drinks per week and/or ≥4 standard drinks per occasion for males and >7 standard drinks per week and/or ≥3 standard drinks per occasion for females. A standard drink is 12 oz of beer (5% alcohol), 5 oz table wine (12% alcohol), or 1.5 oz of spirits (40% alcohol).
* Known or suspected, in the opinion of the Investigator, renal disease or renal impairment.
* Twelve-lead ECG demonstrating a QT interval corrected for heart rate according to Fridericia (QTcF) that is >500 msec or other clinically relevant abnormalities as judged by the Investigator at Screening.
* Use of or intention to use excluded or contraindicated medication(s) or supplements, including any medication known to be a moderate or potent inducer or inhibitor of the cytochrome P450 3A4 enzyme, within 14 days prior to Screening and for the duration of the study.
* Receipt of ≥14 days of systemic immunomodulator therapy (eg, oral corticosteroids) within 3 months of Screening.
* Prior to the first dose of study drug and during study participation, the subject has received any vaccine, investigational agent, or biological product within 30 days or 5 times the half-life, whichever is longer. Note: Influenza vaccination within 7 days of Screening is allowed.
* Use of St John's wort within 28 days prior to the first dose of study drug and for the duration of the study.
* History of or currently experiencing a medical condition or any other finding (including laboratory test results) that, in the opinion of the Investigator, might confound the results of the study; pose an additional risk in administering study drug to the subject; could prevent, limit, or confound the protocol-specified assessments; or deems the subject unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rottinghaus, MD, Study Director — Enanta Pharmaceuticals, Inc
Locations (29):
- United States (12):
  - Central Alabama Research, Birmingham, Alabama
  - Cahaba Research Inc. - Birmingham, Pelham, Alabama
  - Saint Joseph's Clinical Research, Anaheim, California
  - Torrance Clinical Research Institute, Lomita, California
  - Miami Clinical Research - ClinEdge - PPDS, Miami, Florida
  - Pioneer Clinical Research LLC, Bellevue, Nebraska
  - Meridian Clinical Research, Norfolk, Nebraska
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Carolina Research Center, Shelby, North Carolina
  - PMG Research of Wilmington, Wilmington, North Carolina
  - Progressive Medicine of the Triad, LLC, Winston-Salem, North Carolina
  - FMC Science, Lampasas, Texas
- Instituto Medico Platense, Buenos Aires, Argentina
- Bulgaria (6):
  - Diagnostic and Consulting Center Aleksandrovska EOOD, Sofia, Sofia-Grad
  - Medical Center Hera, Sofia, Sofia-Grad
  - Multiprofile Hospital for Active Treatment Puls, Blagoevgrad
  - Specialized Hospital for Active Treatment of Pneumophthisiatric Diseases - Haskovo EOOD, Haskovo
  - Medical Center Zdrave-1 OOD, Kozloduy
  - Medical Center Tara OOD, Veliko Tarnovo
- New Zealand (2):
  - Lakeland Clinical Trials - Waikato, Hamilton
  - Lakeland Clinical Trials, Rotorua
- Poland (2):
  - Alergo-Med Specjalistyczna Przychodnia Lekarska Sp. z.o.o, Tarnów, Lesser Poland Voivodeship
  - Specjalistyczny Osrodek Leczniczo-Badawczy Zbigniew Zegota, Ostróda
- Clinical Projects Research SA pty Ltd, Worcester, Western Cape, South Africa
- Ukraine (5):
  - Communal Non-Profit Enterprise City Clinical Hospital #1 of Ivano-Frankivsk City Council, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Municipal Enterprise The 1st City Clinical Hospital of Poltava City Council, Poltava, Poltava Oblast
  - City Outpatient Clinic #9, Kyiv
  - Medical Center of LLC Preventclinic, Kyiv
  - Limited Liability Company Medical Center Consilium Medical, Kyiv

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EDP-938 | Placebo
Started | 41 | 41
Completed | 31 | 30
Not Completed | 10 | 11

BASELINE CHARACTERISTICS:
Population: The Safety (SAF) population included 81 subjects (98.8% of total randomized subjects) composed of all subjects who received at least one dose of study drug or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | EDP-938 | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (14.61) | 47.8 (14.14) | 47.4 (14.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 15 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 31 | 34 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 3 | 5
  White | 35 | 36 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Symptom Score (TSS) Area Under the Curve (AUC)
Description: Assessed by the RSV Symptom Diary, including 13 items assessing the severity of RSV-related signs and symptoms. The diary uses a 4-point scale that consists of grading symptoms on a scale of 0 to 3 for each item, where Grade 0 is Absent, Grade 1 is Noticeable, Grade 2 is Bothersome but not preventing activity, and Grade 3 is Bothersome and interfering with activities. TSS is derived daily by summing of the 13 observed symptom grade values from Day 1 through Day 14 to generate the curve for analysis.
Time Frame: Day 1 through Day 14
Population: The mITT population included 66 subjects, comprised of all randomized subjects positively diagnosed using the central RT-PCR test who received at least one dose of the assigned study drug or placebo. Per SAP, one subject in the EDP-938 group with only baseline data was excluded from analysis.
Measure: Mean (Standard Deviation); unit: days x Score
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 33 | 33
days x Score
  RSV A: number analyzed (Participants) | 18 | 19
  RSV A | 93.64 (97.180) | 62.53 (40.310)
  RSV B: number analyzed (Participants) | 15 | 14
  RSV B | 73.75 (66.652) | 78.34 (58.051)

2. Secondary Outcome: RSV RNA Viral Load Area Under the Curve (AUC)
Description: RSV RNA viral load as measured in nasopharyngeal swab samples by RT-qPCR on Days 1 (Baseline, time 0), 3, 5, 9, and 14 to generate curve for analysis.
Time Frame: Day 1 through Day 14
Population: The mITT population included 66 subjects, comprised of all randomized subjects positively diagnosed using the central RT-PCR test who received at least one dose of the assigned study drug or placebo. Per SAP, one subject in the placebo group and two subjects in the EDP-938 group with only baseline data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: days x log10 copies/mL
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 31 | 32
days x log10 copies/mL | 37.00 (24.003) | 46.96 (21.002)

3. Secondary Outcome: Number of Subjects With RSV RNA Viral Load Below Limit of Detection (LOD)
Description: Proportion of patients that have undetectable RSV RNA by qRT-PCR at Days 3, 5, 9 and 14.
Time Frame: Days 3, 5, 9 and 14
Population: Based on subjects positively diagnosed using the central RT-PCR test and with detectable viral load at baseline and non-missing viral load assessment at the respective visit and is used as a denominator in the percentage calculation.
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 33 | 33
Participants
  Day 3: number analyzed (Participants) | 30 | 32
  Day 3 | 5 | 2
  Day 5: number analyzed (Participants) | 29 | 30
  Day 5 | 12 | 5
  Day 9: number analyzed (Participants) | 31 | 32
  Day 9 | 15 | 11
  Day 14: number analyzed (Participants) | 31 | 30
  Day 14 | 26 | 23

4. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Day 1 through Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | EDP-938 | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 11 | 11

ADVERSE EVENTS:
Time Frame: Participants were assessed over a period of two weeks; five days of dosing and nine days of follow-up.
Arm/Group | EDP-938 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 11/40 | 11/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EDP-938 (N=40) | Placebo (N=41)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 2 (2)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 1 (1) | 0 (0)
Urine ketone body present (Investigations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04196101/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04196101/SAP_002.pdf